CLINICAL TRIAL: NCT05154435
Title: Comparison of the Effects of Perioperative Targeted and Traditional Fluid Management on Inferior Vena Cava Collapsibility Index and Postoperative Complications in Geriatric Patients Undergoing Proximal Femoral Surgery
Brief Title: the Effects of Perioperative Goal Directed and Conventional Fluid Management on the IVC Collapsibility Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FSMTRH1
Record Dates: First submitted 2021-11-16; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Femoral Neck Fractures
Keywords: intraoperative care, hemodynamic monitoring, fluid therapy
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: A total of 60 patients over the age of 65, who were scheduled for proximal femoral surgery due to intertochanteric fracture, and operated with ASA1-3 risk will be included in the study. The patients will be randomized into two groups as Group K (n=30) and Group H (n=30) by the closed envelope method and the patients will not know their groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients who accepted to participate in the study and the doctor who measured the inferior vena cava did not know the groups of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup HYT (Active Comparator): The group (GRUP HYT) to be treated with targeted fluid therapy will be monitored with a Mostcaretm (Vygon, VytechHealth, Padova, Italy) pulse contour hemodynamic monitor after arterial cannulation. Cardiacindex (CI), stroke volume variance (SVV), pulse pressure variance (PPV), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI), oxygen delivery (Do2), arterial elastance (Ea) measurements and mean arterial pressure Every 5 minutes to be followed, fluid therapy will be planned in accordance with our algorithm.
  Interventions: Drug: mostcare hemodynamic monitor
- Grup KON (No Intervention): Fluid deficit due to fasting time will be calculated in accordance with the 4-2-1 rule for patients in Group KON. half of the calculated fluid volume in the first hour; the remaining half will be given at the 2nd and 3rd Hours. (4ml/kg/hr for the first 10 kilograms, 2ml/kg/hr for the second 10 kg, 1ml/kg/hr for each subsequent kilogram). Maintenance fluid will be considered as a medium-sized surgical trauma and will be given at 4 ml/kg/hr. Hemorrhages will be replaced with 3 times the blood loss with balanced crystalloid or 1 times HES.

INTERVENTIONS:
Drug: mostcare hemodynamic monitor — mostcare hemodynamic monitoring integrated into the radial artery catheter. According to the data obtained, intraoperative fluid management was arranged with certain algorithms.
  Other Names: minimally invasive cardiac output monitors
  Arms: Grup HYT

SUMMARY:
The investigators aimed to compare the effects of targeted fluid management and traditional fluid management on the inferior vena cava collapsibility index in participants who will undergo proximal femoral surgery. In addition, the amount of fluid given, blood products, the number of perioperative hypotensive events, perioperative hemodynamics, perioperative and postoperative blood gas analysis, perioperative urine output and bleeding amount, postoperative complications (cardiac, respiratory, renal, etc.), postoperative 30-day mortality, nausea and vomiting score, It was aimed to evaluate and compare the postoperative hospitalization day as secondary.

DETAILED DESCRIPTION:
Hip fracture surgeries have become one of the most frequently performed surgeries with the increase in the aging population in recent years. Perioperative fluid management of geriatric patients who become prone to dehydration due to malnutrition, decreased functional capacity, impaired cognitive functions after hip fracture development; It is important in terms of reducing complications in the postoperative period and perioperative hemodynamics.

The traditional approach to perioperative fluid administration is the fluid deficit for the fasting period with the '4-2-1' rule (4ml/kg/hr for the first 10 kg, 2ml/kg/hr for the second 10 kg, 1ml/kg/hr for each subsequent kg). ) calculation. The fluid and blood losses in the surgical area and the fluid deficit are estimated and replaced. In order to replace the volume deficit caused by blood loss, crystalloid is used 3 times the amount of bleeding, taking into account the crystalloid movement into the extravascular compartment. Static parameters such as blood pressure, heart rate, and urine volume, which are followed in fluid management with the traditional approach, support the estimation of intravascular volume.

Maintaining intravascular euvolemia throughout the perioperative period is ideal. Both hypovolemia and hypervolemia are associated with increased postoperative morbidity. While vasoconstriction due to hypovolemia, decreased oxygen delivery, decreased tissue perfusion and dysfunction in peripheral organs can be observed; Tissue edema due to hypervolemia, impaired tissue perfusion, local inflammation, delayed wound healing, wound infection and anastomotic leaks can be seen. There is no clear consensus on how to perform optimal fluid management in this population, which has many comorbidities and is at high risk for postoperative complications.

The search for an optimal fluid regimen to avoid excessive intravascular volume overload and maximize tissue perfusion has brought individualized targeted fluid replacement therapies with the help of developing technology. In the targeted therapy (HYT) approach, basic physiological variables related to cardiac output or global O2 distribution are measured with the aim of improving tissue perfusion and clinical outcome. Replacement by crystalloid, colloid or blood products is adjusted according to the dynamic process according to the measured physiological variables. Methods such as pulmonary artery catheter, esophageal doppler, central venous pressure measurement, echocardiography, lactate, central venous saturation, thoracic bioimpedance and arterial waveform analysis can be used to determine physiological targets.

Arterial waveform analysis provides estimation of cardiac output based on continuous analysis of the waveform, a complex physiological signal determined by the interaction of left ventricular stroke volume, systemic vascular resistance, and vascular compliance. Arterial waveform analysis stands out because it can measure continuous cardiac output and does not require a central venous catheter. There are invasive, minimally invasive and non-invasive waveform monitoring systems.

One of the methods used in the evaluation of intravascular volume status is the evaluation of the diameter of the inferior vena cava (IVC) and its collapsibility, which changes with respiration. It can be done at the bedside, it is a fast and noninvasive method.

Inferior vena cava collapsibility index (cIVC) can be used as an indicator of fluid response and a guide in fluid management in critically ill breathing spontaneously.

Several meta-analyses have reported that individualized targeted perioperative fluid managements reduce organ-specific complications in patients undergoing major surgery. In a study, it was stated that targeted fluid therapy in patients with proximal femur fractures decreased the total amount of fluid administered and could reduce postoperative complications.

Although the necessity of providing adequate intravascular volume in perioperative fluid management is obvious, an optimal fluid management guideline has not been established in geriatric and emergency cases with high mortality. The investigators aimed to compare the cIVC measurements and perioperatively administered fluid volumes of the patients who the investigators performed fluid management with the arterial waveform analysis method, which measures the minimally invasive continuous cardiac output, and the patients with whom the investigators had fluid management with traditional methods, and to examine the postoperative effects.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* 1-3 ASA anesthesia risk
* Planned to undergo proximal femoral surgery due to intertochanteric fracture

Exclusion Criteria:

* cardiac arrhythmia,
* chronic renal failure and those on dialysis,
* heart failure,
* aortic insufficiency,
* active lower/upper respiratory tract infections,
* inferior vena cava cannot be clearly visualized by USG, BMI>35, Patients in need of postoperative intensive care or ASA4, Patients with advanced obstructive or restrictive respiratory diseases, Patients under 65 years of age.

Ages: 65 Years to 101 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Inferior vena cava (IVC) collapsibility index | one month
  inspiratory IVC diameter and expiratory IVC diameter will measured and collapsibility index will be calculated

SECONDARY OUTCOMES:
amount of given crystalloid and colloid volume | one month
  Total delivered crystalloid, colloid, urine output, and bleeding volume (ml) will be recorded during the intraoperative period.
arterial blood gas analysis | one month
  preoperative and postoperative hemoglobin, hematocrit, sodium, potassium, lactate, base excess, bicarbonate values will be compared
postoperative complications (yes or no) | one month
  patients before discharge, hemorrhagic, cerebral, infective complications, etc. will be questioned in terms of the presence or absence of complications.
postoperative 30-day mortality (yes or no) | one month
  Postoperative 30-day mortality patients will be called by phone and questioned.

CONTACTS AND LOCATIONS:
Overall Officials: arzu yıldırım ar, ass prof, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes